CLINICAL TRIAL: NCT05216783
Title: Effect of Motivational Interviews on Childbirth Perception and Childbirth Self-Efficacy: A Randomized-Controlled Trial
Brief Title: Effect of Motivational Interviews on Childbirth Perception and Childbirth Self-Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Sümeyye Barut, Lecturer, Inonu University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2019/451
Record Dates: First submitted 2021-12-16; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Trauma; Childbirth; Self Efficacy
Keywords: Childbirth; Motivational Interviewing; Self-Efficacy; Perception; nullipara
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: This study was designed as a randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The Personal Information Form, the Traumatic Childbirth Perception Scale (TCPS), and the short-form Childbirth Self-Efficacy Inventory (CBSEI-32) were utilized for the collection of research data. First of all, the TCPS was applied to the pregnant women, and the pregnant women who obtained a score above 53 points (moderate-level traumatic childbirth perception) from the TCPS were invited to the research. Next, the Personal Information Form and the CBSEI-32 were applied to the pregnant women who agreed to participate in the research. The motivational interviews were held with the pregnant women in the experimental group once a week for four weeks. No initiative was applied to the pregnant women in the control group. The TCPS and CBSEI-32 were applied to all participant pregnant women after four weeks following the first application. The application of the measurement tools took 10-15 minutes.
  Interventions: Behavioral: Motivational Interviews
- Control (No Intervention): The researchers applied no initiative to the control group, and the pregnant women in the control group solely had the routine checks performed at the city hospital. At the end of the study, the questions of pregnant women in the cotrol group about childbirth were answered. Before applying the initiative to the experimental group, the researcher (SB) had had training about motivational interview techniques.

INTERVENTIONS:
Behavioral: Motivational Interviews — The qualitative research studies performed on the traumatic childbirth experiences indicated that the pregnant women's interaction and communication with the midwives were more effective than the medical intervention methods that were applied.
  Arms: Experimental

SUMMARY:
Aim: The aim of this study to determine the effect of motivational interviews on the perception and self-efficacy of birth in nullipars with a perception of traumatic birth.

Materials and Methods: The study was conducted in a randomized controlled, between November 2019 and November 2020 in the obstetrics outpatient clinics of Elazig Fethi Sekin City Hospital. In the power analysis, the sample size was calculated as at least 83 pregnant women for each group (83 experiment, 83 control). Data were collected with Descriptive Information Form, Traumatic Childbirth Perceptions Scale (TCPS) and Childbirth of Self-Efficacy Scale-Short From (CBSE). Pregnant women in the experimental group were held with four sessions of motivational interviews one week a part. No intervention was made for the pregnant women in the control group. Descriptive statistics, chi-square test, t test for dependent and independent groups were used in data analysis

DETAILED DESCRIPTION:
Materials and Methods

Research Design and Sample

This study was designed as a randomized controlled trial in which the research subjects were randomly assigned to an experimental group that took part in the motivational interview and a control group. The research population was comprised of nulliparous women who were admitted to the obstetrics polyclinic in a city hospital in Turkey. Only a city hospital and a university hospital were located in the province center where the research took place. Mostly, the high-risk pregnancies are followed up in the university hospital. Therefore, the research was conducted in the city hospital. According to the records of the city hospital, 6,768 pregnant women were admitted to the obstetrics polyclinic in 2019. The research data were collected from July 2019 to November 2020.

Web-based sample size calculation was used in calculating the sample size for the research. As per the power analysis conducted with a 5% margin of error, 95% confidence interval at two-tailed statistical significance level, and 80% power, the sample size was calculated as 83 pregnant women for each group (83 pregnant women for the experimental group, 83 pregnant women for the control group) assuming that the mean Traumatic Childbirth Perception Scale score that was 70.57±21.89 points before applying the motivational interviews (Aktaş, 2018) would go down by 9 points following the motivational interviews. The process of sample selection took place in conformity with the criteria prescribed by the Consolidated Standards of Reporting Trials (CONSORT).

The criteria for being included in the research were as follows: (1) having the ability to communicate, (2) being within 28-36 weeks of pregnancy, (3) being aged 18 or above, (4) having a live singleton fetus, (5) having no pregnancy-related risk (pre-eclampsia, diabetes, cardiac disease, placenta previa, oligohydramnios, and so on), (6) having no problem about the fetus's health (fetal anomaly, intrauterine growth restriction, and so on), (7) having a medium or a higher level of traumatic childbirth perception according to the Traumatic Childbirth Perception Scale (≥53 points). The criterion for being excluded from the research was to have a condition that would prevent the woman from having a normal birth (total placenta previa and so on).

The pregnant women who satisfied the inclusion criteria stipulated for the research were assigned to the experimental group (n=107) and control group (n=100) through simple randomization according to the historical order of their admittance to the polyclinic. Out of 107 pregnant women included in the experimental group, 13 women were excluded from the research after the first motivational interview (two pregnant women for being diagnosed with a high-risk pregnancy, three pregnant women for having a premature birth, and eight women for not attending the research), 8 women were excluded from the research after the second motivational interview (two pregnant women for being diagnosed with a high-risk pregnancy, two pregnant women for having a premature birth, and four women for not continuing to attend the research), and 3 women were excluded from the research after the third motivational interview (three pregnant women for having a premature birth). Of 100 pregnant women included in the control group, 17 women were excluded from the research after the first meeting with the researcher (four pregnant women for being diagnosed with a high-risk pregnancy, six pregnant women for having a premature birth, and seven women for not attending the research). Thus, the research was finalized with the participation of 166 pregnant women in total (83 pregnant women in the experimental group, 83 pregnant women in the control group.

Data Collection Tools The Personal Information Form, the Traumatic Childbirth Perception Scale (TCPS), and the short-form Childbirth Self-Efficacy Inventory (CBSEI-32) were utilized for the collection of research data.

Personal Information Form

The Personal Information Form was created by the researchers upon the review of the relevant literature. The questions in the form pertained to the participant woman's sociodemographic characteristics (age, education level, employment status, income level, and so on) and data about her pregnancy (how many pregnancies the woman had, whether the current pregnancy was desired by the woman, and so on).

Traumatic Childbirth Perception Scale (TCPS)

Yalnız et al. (2016) developed the scale to evaluate the traumatic childbirth perception levels of the women at reproductive age and performed the validity and reliability test for the scale in Turkish. The scale has a total of 13 questions that cover thoughts and emotions such as anxiety, fear, and worry felt by the women while thinking about the concept of childbirth. Each question is scored from 0 (I am not afraid at all) to 10 points (I am very afraid). The mean of scores obtained from the scale indicates the traumatic childbirth perception level. The minimum and maximum scores to be obtained from the scale are successively 0 and 130 points. A high score obtained from the scale demonstrates that the pregnant woman has high-level traumatic childbirth perception. The scores ranging from 0 to 26, from 27 to 52, from 53 to 78, from 79 to 104, and from 105 to 130 consecutively refer to very low, low, moderate, high, and very high levels of traumatic childbirth perception. The Cronbach's alpha coefficient was calculated as 0.89 for the scale. Under this study, it was found as 0.82 for the scale.

Short-Form Childbirth Self-Efficacy Inventory (CBSEI-32)

The inventory was developed by Ip et al. in 2005 to measure the women's levels of self-efficacy in childbirth and the validity and reliability test for the inventory was performed in Turkish in 201. It has two factors, that is, outcome expectancy (OE-16) and efficacy expectancy (EE-16), and each factor has 16 questions. The minimum and maximum scores to be obtained from each factor are successively 16 and 160 points. A high score to be obtained from each factor shows that the pregnant woman has high-level efficacy and outcome expectancy in relation to the act of giving birth. In this Likert-type inventory, the answers given to the questions are scored from 1 to 10 points. The respondent choices are expressed as 'not at all helpful' (1 point) and 'very helpful' (10 points) for each question under the OE-16 whilst they are expressed as 'very sure' (1 point) and 'not at all sure' (10 points) in the first thirteenth questions and as 'not at all sure' (1 point) and 'very sure' (10 points) in the questions 14-16 under the EE-16. The first 13 questions in the EE-16 are reverse-scored. The minimum and maximum total scores to be obtained from the inventory are respectively 32 and 320 points. A high score to be obtained from the inventory indicates that the pregnant woman has high-level self-efficacy in childbirth. The Cronbach's alpha coefficient was calculated as 0.90 for the inventory. Under this study, it was found as 0.92 for the inventory.

Data Collection

The research data were collected by the researchers through the face-to-face interview method in the school of pregnant women located in the city hospital. First of all, the TCPS was applied to the pregnant women, and the pregnant women who obtained a score above 53 points (moderate-level traumatic childbirth perception) from the TCPS were invited to the research. Next, the Personal Information Form and the CBSEI-32 were applied to the pregnant women who agreed to participate in the research. The motivational interviews were held with the pregnant women in the experimental group once a week for four weeks. No initiative was applied to the pregnant women in the control group. The TCPS and CBSEI-32 were applied to all participant pregnant women after four weeks following the first application. The application of the measurement tools took 10-15 minutes.

Intervention

The researcher (SB) had motivational interviews with the pregnant women in the experimental group once a week for four weeks in the research. The aim of motivational interviews is to enable that pregnant women understand the traumatic childbirth perception, take action for change, and believe in change. The interview sessions were held with the pregnant women in the experimental group on an individual basis in the school of pregnant women of the city hospital. Each motivational interview session lasted 15-30 minutes on average. During the interviews, the consultancy service on the birth-related topics (what the traumatic childbirth perception is, childbirth fear and its effects, procedures performed in the delivery room, delivery process, initiatives to be taken to mitigate the traumatic childbirth experience during delivery, and so on) was offered to change the pregnant women's negative childbirth perceptions and enhance their childbirth self-efficacy. The researchers applied no initiative to the control group, and the pregnant women in the control group solely had the routine checks performed at the city hospital. At the end of the study, the questions of pregnant women in the cotrol group about childbirth were answered. Before applying the initiative to the experimental group, the researcher (SB) had had training about motivational interview techniques.

Statistical Analysis

The statistical analysis of the data obtained from the research was conducted with SPSS (Statistical Package for Social Science) 20.0. In the research, the numerical data were expressed as the means and standard deviations while the nominal data were indicated in frequencies and percentages. The chi-squared test was used in the inter-group comparison of the nominal data. In the evaluation of numerical data, firstly, the Kolmogorov-Smirnov test was utilized to identify whether the data had a normal distribution. As the research data were normally distributed, the independent samples t-test was used in the comparison of two groups whilst the dependent samples t-test was employed in the intra-group comparison. Statistical significance was identified if the P-value was lower than 0.05 (p<0.05).

ELIGIBILITY:
Inclusion Criteria:

* having the ability to communicate,
* being within 28-36 weeks of pregnancy,
* being aged 18 or above,
* having a live singleton fetus,
* having no pregnancy-related risk (pre-eclampsia, diabetes, cardiac disease, placenta previa, oligohydramnios, and so on),
* having no problem about the fetus's health (fetal anomaly, intrauterine growth restriction, and so on),
* having a medium or a higher level of traumatic childbirth perception according to the Traumatic Childbirth Perception Scale (≥53 points).

Exclusion Criteria:

* The criterion for being excluded from the research was to have a condition that would prevent the woman from having a normal birth

Ages: 28 Weeks to 36 Weeks | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Nullipars woman
Enrollment: 166 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-02-12 (Actual)

PRIMARY OUTCOMES:
Traumatic Childbirth Perception Scale (TCPS) | Change from Traumatic Childbirth Perception at 4 weeks
  It is used to evaluate the traumatic childbirth perception levels of the women at reproductive age. The scale has a total of 13 questions that cover thoughts and emotions such as anxiety, fear, and worry felt by the women while thinking about the concept of childbirth. Each question is scored from 0 (I am not afraid at all) to 10 points (I am very afraid). The mean of scores obtained from the scale indicates the traumatic childbirth perception level. The minimum and maximum scores to be obtained from the scale are successively 0 and 130 points. A high score obtained from the scale demonstrates that the pregnant woman has high-level traumatic childbirth perception. The scores ranging from 0 to 26, from 27 to 52, from 53 to 78, from 79 to 104, and from 105 to 130 consecutively refer to very low, low, moderate, high, and very high levels of traumatic childbirth perception

SECONDARY OUTCOMES:
Short-Form Childbirth Self-Efficacy Inventory (CBSEI-32) | Change from Short-Form Childbirth Self-Efficacy at 4 weeks
  It has two factors, that is, outcome expectancy (OE-16) and efficacy expectancy (EE-16). The minimum and maximum scores to be obtained from each factor are successively 16 and 160 points. A high score to be obtained from each factor shows that the pregnant woman has high-level efficacy and outcome expectancy in relation to the act of giving birth. The minimum and maximum total scores to be obtained from the inventory are respectively 32 and 320 points. A high score to be obtained from the inventory indicates that the pregnant woman has high-level self-efficacy in childbirth.

CONTACTS AND LOCATIONS:
Overall Officials: Sümeyye barut, PhD, Principal Investigator — Firat University
Locations (1):
- Fırat University, Elâzığ, Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No